CLINICAL TRIAL: NCT06696222
Title: Fermented Vegan Optimized Diet in Health and Colitis
Acronym: FAVORIT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Region Skane (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 2024-05870 FAVORIT
Record Dates: First submitted 2024-11-11; First posted 2024-11-20 (Actual); Last update posted 2025-07-01 (Actual); Status verified 2025-06

CONDITIONS: Healthy Volunteers; Inflammatory Bowel Disease (IBD)
Keywords: diet; ulcerative colitis; Crohn's disease; vegetarian diet
MeSH Terms: conditions — Inflammatory Bowel Diseases; Colitis, Ulcerative

STUDY DESIGN:
Intervention Model Description: Prospective non-randomized intevention study where everyone serves as their own control
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Vegetarian yogurt alternative (Active Comparator): Participants will consume vegatarian based alternatives instead of ordinary yogurt.
  Interventions: Dietary Supplement: Vegetarian yogurt
- Placebo: Ordinary yogurt based diet (Placebo Comparator): Participants will consume regular yogurt.
  Interventions: Dietary Supplement: Placebo
- Vegetarian meat alternative (Active Comparator): The participants will consume a vegetarian alternative to meat.
  Interventions: Dietary Supplement: Vegetarian meat alternative
- Placebo - ordinary meat diet (Placebo Comparator): The participants will consume an ordinary meat based diet.
  Interventions: Dietary Supplement: Ordinary meat diet

INTERVENTIONS:
Dietary Supplement: Vegetarian yogurt — Vegetarian yogurt alternative will be uesd.
  Arms: Vegetarian yogurt alternative
Dietary Supplement: Placebo — Ordinary diet with dairy based yogurt
  Arms: Placebo: Ordinary yogurt based diet
Dietary Supplement: Vegetarian meat alternative — Vegetarian meat alternative consumed
  Arms: Vegetarian meat alternative
Dietary Supplement: Ordinary meat diet — Ordinary meat diet used as placebo
  Arms: Placebo - ordinary meat diet

SUMMARY:
The diet is assumed to contribute to many of our present non-communicable diseases. Vegetarian products are instead considered to be health promoting, However, it is not verified that the modern vegetarian and vegan products are healthier than the ones they are meant to replace. Products based on vegetables are nowadays often produced with advanced techniques and can therefore differ substantially from the original vegetables.

The epithelium in the gut is protected by a mucus layer that efficiently prevents bacteria to encounter the epithelium and even to translocate into the gut and the blood stream. In several inflammatory conditions such as e.g., inflammatory bowel disease (IBD) the barrier integrity is disrupted, and translocation will occur. Fibers are important for the gut microbiota enabling the production of short chain fatty acids (SCFA) that is necessary as nutrition for the epithelial cells, Fibers also promote the development of mucus.

The aim of the present study is to evaluate components in the diet that is claimed to be health promoting even though they sometimes can be a hazard to your health. Both fibers and antinutrients can be found in these dietary regimens. The health effects of these products will be studied by analysis of the gut microbiota and the barrier integrity as markers of the health status. Gut microbiota will be analyzed with next generation sequencing and q-PCR (polymerase chain reaction). Diversity and the occurrence of different species will be determined. The barrier integrity will be estimated by analysis of bacterial DNA in blood and presence of live bacteria.

The study consists of two different parts:

1a. 60 health volunteers are divided into two groups. One group consumes ordinary dairy based yogurt and the other a yogurt based on vegan products for four weeks to enable a change in the gut microbiota. At start and after four weeks fecal samples and questionnaires about the general health and gastrointestinal symptoms will be retrieved. It should be noted that the compounds offered can be bought in the ordinary shops.

1. b. The same design as above but with IBD patients instead. Their disease activity will be monitored by scoring sheets and regular blood tests as a part of their regular check-up.
2. a. The same design as in 1a but with comparison between a regular meat-based diet and a diet with vegetarian meat substitutes instead.

2b. The same design as I 2a but with IBD patients. Healthy volunteers will be invited wit advertisements. The IBD patients will be recruited at the out-patient clinic at the Dept of Gastroenterology at Skåne university hospital, Sweden. Before inclusion their disease activity will be monitored.

The study is a prospective non-randomized intervention study including both men and women. Each individual will serve as their own control. The meals based on meat substitutes will be composed in cooperation with a dietitian. The estimated amount of yogurt is 200-250 gram/day, and the amount of meat is 150-200 gram/day.

DETAILED DESCRIPTION:
The present dietary habits in the western world result in ill health in the community. The diet is assumed to contribute to many of the non-communicable auto-inflammatory diseases we suffer from today. For example, in 2019 excess caloric intake, insufficient consumption of whole grains and vegetables, and overexaggerated intake of meat and salt were considered to contribute to the disease burden. Processed food with a lot of salt, sugar and emulsifying agents are considered extra harmful.

A diet instead predominantly consisting of vegetarian products is considered to be health promoting, However, it is not verified that the modern vegetarian and vegan products are healthier than the ones they are meant to replace. Products based on vegetables are nowadays often processed with advanced techniques and can therefore differ substantially from the original vegetables that are used. It is therefore indicated to evaluate their putative health promting effects.

The epithelium in the gut is protected by a mucus layer that efficiently prevents bacteria to encounter the epithelium and even to translocate into the gut and in the next step the blood stream. In several inflammatory conditions such as e.g., inflammatory bowel disease (IBD), i.e., ulcerative colitis and Crohn's disease, the barrier integrity is disrupted, and translocation may occur. Fibers are considered important for the gut microbiota enabling the production of short chain fatty acids (SCFA) that is necessary as nutrition for the epithelial cells, Fibers also promote the development of mucus.

The aim of the present study is to evaluate components in the diet that are claimed to be health promoting even though they sometimes can be a hazard to your health instead. Both fibers and antinutrients can be found in these dietary regimens. The health effects of these products will be studied by analysis of the gut microbiota and the barrier integrity as markers of the health status. Gut microbiota will be analyzed with next generation sequencing and q-PCR (polymerase chain reaction). Diversity and the occurrence of different species will be determined. The barrier integrity will be estimated by analysis of bacterial DNA in blood and in some cases also presence of live bacteria.

The study consists of two different parts:

1a. 60 health volunteers are divided into two groups. One group consumes ordinary dairy based yogurt and the other a yogurt based on vegan products (from the same company and with the same bacterial composition). The duration is four weeks to enable a change in the gut microbiota. Fecal samples will be collected at start and after four weeks. They will also respond to questionnaires about their general well-being and if any gastrointestinal complaints should occur. It should be noted that the compounds are already used by consumers and can be bought in the ordinary shops.

1. b. The same design as above but with IBD patients instead. Their disease activity will be monitored by scoring sheets and regular blood tests as a part of their regular check-up.
2. a. The same design as in 1a but with comparison between a regular meat based diet and a diet with vegetarian meat substitutes instead.

2b. The same design as I 2a but with IBD patients.

Healthy volunteers will be invited wit advertisements. The IBD patients will be recruited at the out-patient clinic at the Dept of Gastroenterology and Nutrition at Skåne university hospital. Before inclusion their disease activity will br monitored according to established principles.

The study is a prospective non-randomized intervention study including both men and women. Each individual will serve as their own control. The meals based on meat substitutes will be composed in cooperation with a dietitian. The estimated amount of yogurt is 200-250 gram/day, and the amount of meat is 150-200 gram/day. These amounts is based on what is recommended as a daily intake.

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteers in two groups
* IBD in two groups (ulcerative colitis or Crohn's disease)

Exclusion Criteria:

* For healthy any disease requiring medication
* For IBD previous extensive operation
* For both antibiotics the past month

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 240 (Estimated)
Dates: Start 2024-11-18 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Diversity and microbial composition | Four weeks
  Gut microbiota will be analyzed at start and after four weeks. The health promoting efect of the diet will be estimated with analysis of the alfa and beta diversity as well as microbila composition down to species level to determine the balance betweedn beneficial and harmful species. Based on the complexity of the micorbiota it is not possible to state any specific value that should be achieved.

SECONDARY OUTCOMES:
Barrier integrity | Four weeks
  The barrier function will be estimated by analysing the presence of bacterial DNA in blood. The health promoting effect of the diet on barrier integrity will be estimated with analysis of the amount of bacterial DNA in the blood stream. Since this ia a study investigating new findings based on one previous article it is not possible to state any specific cut-off value. .

CONTACTS AND LOCATIONS:
Overall Officials: Klas Sjöberg, Adj prof, Principal Investigator — Dept of Gastroenterology
Locations (1):
- Dept of Gastroenterology, Malmo, Sweden

IPD SHARING:
Plan to Share IPD: Yes
Data on group level can be shared upon request.
Supporting Information: Study Protocol, CSR
Time Frame: Dcember 31, 2026 until December 31, 2027
Access Criteria: In order to establish research cooperation.